CLINICAL TRIAL: NCT06764550
Title: Molecular and Microbiota Signatures Underlying Colonic Diverticular Disease - Caratterizzazione Dei Meccanismi Molecolari e Del Microbiota Nella Malattia Diverticolare Del Colon
Brief Title: Molecular and Microbiota Signatures Underlying Colonic Diverticular Disease
Acronym: GR-Barbaro
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: GR-Barbaro; GR-2018-12367062 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-11

CONDITIONS: Diverticular Disease of Colon
MeSH Terms: conditions — Diverticulosis, Colonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Colonic biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy subjects: Subjects who are asymptomatic for digestive symptoms and without diverticula.
  Interventions: Other: This is an observational study, participants are not assigned an intervention as part of the study.
- Patients with diverticulosis: Patients with diverticula and without symptoms.
  Interventions: Other: This is an observational study, participants are not assigned an intervention as part of the study.
- Patients with symptomatic uncomplicated diverticular disease: Patients with diverticula and with symptoms.
  Interventions: Other: This is an observational study, participants are not assigned an intervention as part of the study.

INTERVENTIONS:
Other: This is an observational study, participants are not assigned an intervention as part of the study. — This is an observational study, participants are not assigned an intervention as part of the study.

SUMMARY:
The pathogenesis of diverticular disease is likely multifactorial in origin. This project aims to study the involvement of environmental factors in the pathophysiology of diverticular disease, the underlying molecular mechanisms, and alterations in the microbiota.

DETAILED DESCRIPTION:
The pathogenesis of diverticular disease is likely multifactorial in origin. Some studies have demonstrated the role of genetic factors, while others have highlighted the role of environmental factors. The present project aims to study the involvement of environmental factors in the pathophysiology of diverticular disease, the underlying molecular mechanisms, and alterations in the microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years.
* Belonging to one of the following groups:

  1. Patients with diverticula of the colon without symptoms.
  2. Patients symptomatic for diverticular disease.
  3. Subjects undergoing colonoscopy for colorectal cancer prevention or follow-up of previous polypectomies, asymptomatic for digestive symptoms.
* Obtaining informed consent.

Exclusion Criteria:

* Acute complicated diverticulitis (bleeding, perforation)
* Previous colon surgery
* Antibiotics or laxatives within the past 90 days
* Pregnancy and/or lactation
* Systemic and psychiatric disorders
* Asthma, food allergies and other allergic-type disorders
* Possible diseases leading to intestinal bacterial contamination (diabetes, blind loop syndrome, rheumatologic diseases).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were recruited from the endoscopy room.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Assess the interaction between host factors and gut microbiota | 3 years
  Assess the interaction between host factors and gut microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Maria Raffaella Barbaro, Biologist, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No